CLINICAL TRIAL: NCT06293209
Title: Effect of Cool Spray and Cold Packs in Reducing Preoperative Edema and Pain in Ankle Fractures in Ubonratchathani: 3-arm Parallel-group RCT
Brief Title: Effect of Cool Spray and Cold Packs in Reducing Preoperative Edema and Pain in Ankle Fractures in Ubonratchathani
Acronym: 3-armRCT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Thai Traditional Medical Knowledge Fund (Other Government)
Responsible Party: Principal Investigator, Watcharachai Potad, MD, Resident of Orthopedics Sunpasitthiprasong hospital, Ubonratchathani, Thailand, Thai Traditional Medical Knowledge Fund
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Sunpasitthiprasong Hospital; Sunpasitthiprasong Hospital (Other: Sunpasitthiprasong Hospital)
Record Dates: First submitted 2024-02-19; First posted 2024-03-05 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-02

CONDITIONS: Ankle Fractures; Swelling; Cryotherapy Effect
MeSH Terms: conditions — Ankle Fractures

STUDY DESIGN:
Intervention Model Description: Population
  The sample group comprises 30 patients admitted for treatment in the male orthopedic surgery department, female orthopedic surgery department, and accident orthopedic surgery department at Sunpasitthiprasong Hospital, Ubon Ratchathani from August 2023 to January 2024. .
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- The control group (non-cryotherapy group) (Placebo Comparator): Routine preoperative protocol ankle fracture on short leg slab compression with bandage
  Interventions: Device: Placebo
- The cold pack group (Active Comparator): The cold pack group consists of patients with ankle fractures who receive cold therapy using ice packs sized 20x20 centimeters. The ice packs are placed in the freezer compartment for 30 seconds after they have solidified, then applied to the injured ankle for 10 minutes, followed by a 10-minute break. This process is repeated every 2 hours for a total of 6 times (from 8:00 AM to 6:00 PM).
  Interventions: Device: 3M cold pack
- The cold spray (Active Comparator): The cold spray group consists of patients with ankle fractures who receive cold therapy using Perskindol cold spray containing Levomenthol. The spray is applied to the injured ankle 5-6 times, followed by a 10-minute break. This process is repeated every 2 hours for a total of 6 times (from 8:00 AM to 6:00 PM).
  Interventions: Device: Perskindol cold spray

INTERVENTIONS:
Device: 3M cold pack — 3M cold pack
  Other Names: cold pack
  Arms: The cold pack group
Device: Perskindol cold spray — Perskindol cold spray
  Other Names: cold spray
  Arms: The cold spray
Device: Placebo — Placebo
  Other Names: non-cryotherapy treatment
  Arms: The control group (non-cryotherapy group)

SUMMARY:
The use of evaporative coolants in the management of acute musculoskeletal injury has received increasing attention recently. However, its efficacy compared with conventional cryotherapy in treating injured human subjects remains unclear.

The purpose of this study is to compare the efficacy of evaporative coolants with that of ice packs in the preoperative management of edema and pain in patients with an ankle fracture

DETAILED DESCRIPTION:
Fractures of the ankle bone are one of the common types of bone fractures found in the general population, accounting for approximately 14% of all fractures They are often found in middle-aged males aged 15-24 years who engage in high-impact physical activities such as sports or high-intensity exercise. They are also found in elderly females with osteoporosis aged 75-84 years The incidence of ankle fractures is 187 per 100,000 population per year Ankle bone fractures usually occur due to excessive force or weight bearing. The main causes of ankle bone fractures can be categorized into three age groups: falls account for up to 61% in the elderly population, sports injuries or repetitive movements in sports or exercises can lead to pain, swelling, and bruising around the ankle joint, or the ankle may appear deformed, which is commonly found in younger age groups, accounting for 22%, and accidents from motor vehicle collisions account for 17% Unimalleolar ankle fractures are the most common type, accounting for 70% of all ankle fractures. Bimalleolar fractures account for approximately 20%, while trimalleolar fractures account for about 7% of all ankle fractures Initial management of ankle injuries involves using the RICE approach, which includes applying ice (I = ice) to the injured area. Cooling the skin with ice packs is a widely used traditional method of caring for injured patients. It has been found that when the skin temperature of bruised areas is reduced below 13.6 degrees Celsius with ice packs, swelling and pain in ankle injuries can be effectively reduced Prolonged use of ice packs for more than 6 days after injury can delay surgery and accelerate tissue recovery after surgery Additionally, studies comparing the effectiveness of reducing swelling in ankle tissue injuries with cold spray and ice packs have found that cold spray is 2-3 times more effective than ice packs in reducing swelling and pain in patients with ankle fractures both before and after surgery However, there has been no study in Thailand on effective cooling methods to reduce swelling and alleviate pain in ankle fractures. Therefore, this research aims to compare the effectiveness of using ice packs and cold spray in reducing swelling and pain before surgery in patients with ankle fractures treated at Sunpasitthiprasong Hospital, Ubon Ratchathani. It is hypothesized that cooling with ice packs and cold spray is effective in reducing swelling and pain in patients with ankle fractures before surgery, and that the effectiveness of ice packs and cold spray in reducing swelling and pain in patients with ankle fractures before surgery differs. This study aims to provide data for developing effective methods and guidelines to reduce swelling and pain in patients with ankle fractures before surgery and may be applied as an alternative option to reduce swelling and pain in patients with fractures in other parts of the body.

ELIGIBILITY:
Inclusion Criteria:

* Thai male and female individuals
* aged 18 years or older.
* diagnosed by the researcher as having unimalleolar fracture, bimalleolar fracture, or trimalleolar fracture requiring surgery.
* capable of reading and writing in the Thai language.

Exclusion Criteria:

* - Fractures in both ankles.
* Pathologic fractures of the ankle bones.
* Simultaneous fractures of the ankle and leg bones.
* Previous history of ankle fractures.
* Nerve-related disorders causing inflammation around the ankle.
* Peripheral artery disease causing blockages in the leg arteries.
* Infections in the ankle area.
* Cold allergy.
* Inability to read and write in the Thai language

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2024-02-28 (Estimated); Study Completion 2024-05-28 (Estimated)

PRIMARY OUTCOMES:
swelling | 5 day before surgery
  Measuring ankle swelling using the figure-of-eight-20 method, which involves measuring the circumference of the ankle and foot using a tape measure placed along the sides of the foot, passing through specific points,3 time and then averaging the measurements obtained in millimeters.

SECONDARY OUTCOMES:
pain score | 48 hours
  Assessing pain levels using the Visual Analog Scale (VAS), a 10-centimeter horizontal line labeled with "no pain at all" at one end and "unbearable pain" at the other. Participants mark their pain level on the scale from 0 to 10, and pain severity is categorized into 5 levels: no pain (0 points), mild pain (1-3 points), moderate pain (4-6 points), severe pain (7-9 points), and extreme pain (10 points).

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Orthopedics, Sunpasitthiprasong hospital, Ubonratchathani, Thailand., Multiple Locations, Ubonrachathani, Thailand

IPD SHARING:
Plan to Share IPD: No